CLINICAL TRIAL: NCT00176189
Title: Clinical Performance of Extended All-Ceramic Fixed Partial Dentures Based on Zircon-Oxide Ceramics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cercon-giant
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-09-26 (Estimated); Status verified 2006-09

CONDITIONS: Tooth Loss, Teeth Replaced Using All Ceramic FPDs
Keywords: FPD, all-ceramic
MeSH Terms: conditions — Tooth Loss

INTERVENTIONS:
Device: All ceramic FPDs

SUMMARY:
Fixed-partial dentures fabricated of zircon-oxide ceramics were introduced in dentistry some time ago. However, the survival rate of all-ceramic extended (up to 47mm) fixed-partial dentures is unknown.

The hypothesis was that long FDPs fabricated of zirkon-oxide withstand masticatory forces in the posterior and anterior regio of the jaw.

DETAILED DESCRIPTION:
30 patients with at least 2 missing posterior or anterior teeth will be included in the study. All patients will receive all-ceramic fixed partial dentures.

ELIGIBILITY:
Inclusion Criteria:

* All patients older 18 years
* At least two missing posterior teeth
* Tooth wear<3

Exclusion Criteria:

* Bruxism
* Mental disorders
* Pregnancy
* Tooth mobility>1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-02; Study Completion 2006-12

PRIMARY OUTCOMES:
Survival rate of the FPDs

SECONDARY OUTCOMES:
Esthetical and functional performance of the FPDs

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rammelsberg, Prof. Dr., Principal Investigator — Department of prosthodontics, University of Heidelberg
Locations (1):
- University of Heidelberg, Heidelberg, Germany